CLINICAL TRIAL: NCT03397524
Title: Tailored Drug Titration Through Artificial Intelligence: an Interventional Study
Brief Title: Tailored Drug Titration Through Artificial Intelligence
Acronym: ARTERY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was dependent on an IT interoperability component requiring additional development.
Sponsor: Optima Integrated Health (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-21426
Record Dates: First submitted 2018-01-05; First posted 2018-01-12 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The interventional arm outcomes will be compared to the control.
Who Masked: Participant
Masking Description: The patient participant will be unaware of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optima4BP (Experimental): optima4BP will receive several types of data to personalize the participant's medication treatment. The data include: remotely measured blood pressure (BP), and information on current medication treatment as well as health updates posted in Epic Electronic Record.
  Interventions: Other: optima4BP
- Standard of Care (No Intervention): The participants randomized to the Standard of Care will follow usual care, as currently followed at the University of California San Francisco.

INTERVENTIONS:
Other: optima4BP — optima4BP will provide the treating physician with a treatment action recommendation for consideration.
  Arms: optima4BP

SUMMARY:
ARTERY is a randomized clinical trial that investigates the benefit of a predictive modeling artificial intelligence in improving the management of anti-hypertensive medication treatment.

DETAILED DESCRIPTION:
The goal of the proposed research is to test a connected medication management platform technology to address medication optimization and non-adherence in chronic disease management. Chronic diseases (such as hypertension, heart failure, diabetes, coronary disease, etc.) are the main causes of morbidity, mortality and healthcare expense in the United States. Poor medication adherence and mismatches in the treatment (due to patient's reported side effect, complexity of treatment, and suboptimal efficacy of a chosen pharmacological treatment) are a major reason of failure in the management of chronic disease. The platform tested in this award will evaluate a complex machine-learning algorithm in treatment optimization for one of the chronic conditions, namely hypertension. The results of the proposed randomized clinical trial, if successful, will lead to a change in the treatment paradigm for chronic diseases. The principal investigator has just completed a pilot study in conjunction with Optima Inrwgrated Health, Inc. (i.e. PRECISION) to successfully test the medication management platform technology and its integration with the electronic medical record (EPIC® platform).

Optima-for-Blood Pressure (O4BP) is a cloud-based artificial intelligence clinical decision support system (CDSS) that evaluates patient status updates in real-time to provide advanced decision recommendations for medication treatment changes, when needed, personalized to each patient. O4BP provides a multiparameter (age, gender, ethnicity, current treatment, comorbidities, side-effects, laboratory values, compliance) overall score computation that ranks possible treatment changes in order of % improvement over current treatment. The goal of the study is to test if blood pressure management by using the O4BP CDSS is superior to standard of care (SOC) (i.e. blood pressure management during office visits).

ELIGIBILITY:
Inclusion Criteria:

* Two or more blood pressure readings of ≥ 150/95 mmHg during primary care office visits in the Department of General Medicine within the last 6 months
* Therapy with medications from at least 1 anti-hypertensive pharmacological agents at the time of the last office visit
* At least minimally "tech-savvy" defined as Ownership of a compatible smartphone Ability to access the internet

Exclusion Criteria:

* Inability to operate a blood pressure cuff
* Incompatible smartphone device (Galaxy S5 Android 5.0)
* Less than minimally "tech-savvy," defined as inability to use the Internet
* Non-compliance with medical follow-up (frequent "no shows")
* Planned coronary revascularization in the next 12 months
* Myocardial infarction, coronary revascularization, stroke, cardiac or aortic surgery in the previous 90 days
* GFR < 30 (CKD stage IV/ V)
* Primary care provider rules out the patient due to comorbidities or other factors

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in systolic BP [SBP] (mmHg) measure in the office | 12 months
  optima4BP leads >6 mmHg of the BP reduction compared to Standard of Care

SECONDARY OUTCOMES:
Reduction in systolic BP [SBP] (mmHg) measure remotely [home monitoring] | 12 months
  optima4BP leads >6 mmHg of the BP reduction compared to Standard of Care baseline through 12 months of enrollment.
Incidence of Adverse Events | 12 months
  Frequency and severity of adverse events (AEs) between baseline and the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Voskerician, Principal Investigator — Optima Integrated Health
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
The patient data will not be shared with other researchers. However, study outcomes will be published in peer-reviewed journals.